CLINICAL TRIAL: NCT05006053
Title: A Qualitative Study of Healthcare Professionals' Perceptions About a Digitally Mediated Intervention for Young People Who Have Experienced Online Sexual Abuse and Its Integration Into Existing NHS and E-therapy Infrastructure
Brief Title: i-Minds Professional Stakeholders Qualitative Study
Status: Completed | Type: Observational
Sponsor: Sandra Bucci (Other)
Collaborators: University of Edinburgh (Other); Greater Manchester Mental Health NHS Foundation Trust (Other); NHS Lothian (Other Government); Pennine Care NHS Foundation Trust (Other Government); Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor-Investigator, Sandra Bucci, Professor, University of Manchester
Organization: University of Manchester (Other)
Other Study IDs: NIHR131848
Record Dates: First submitted 2021-07-29; First posted 2021-08-16 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Child Sexual Abuse, Confirmed, Sequela
MeSH Terms: interventions — Interviews as Topic; Focus Groups

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Qualitative study with healthcare professionals: Healthcare professionals working in Child and Adolescent Mental Health Services, Sexual Assault Referral Centres or with e-therapy providers
  Interventions: Other: Interviews/Focus groups

INTERVENTIONS:
Other: Interviews/Focus groups — Qualitative study (no intervention delivered)
  Other Names: Qualitative Interviews / Focus Groups

SUMMARY:
The main aim of this study is to understand healthcare professionals' perceptions, as well as the barriers and enablers (and unintended consequences), relevant to the uptake of the digital intervention and its future integration into existing NHS infrastructure. We will use a qualitative study design and utilise semi-structured interviews and focus groups to gather the views and opinions from up to 30 healthcare professionals who work with young people to provide mental health and / or sexual assault care across two sites: Greater Manchester, UK and Edinburgh, Scotland.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be up to 30 healthcare professionals who work within NHS services that provide mental health and / or sexual assault support to young people (for example, Child and Adolescent Mental Health Services (CAMHS) and Sexual Assault Referral Centres (SARC)) or organisations that provide digital mental health support to young people (e.g. Kooth).

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Healthcare professionals who work within NHS services in Greater Manchester and Edinburgh that provide mental health and / or sexual assault support to young people (for example, Child and Adolescent Mental Health Services (CAMHS) and Sexual Assault Referral Centres (SARC)) or organisations that provide digital mental health support nationwide to young people (e.g. Kooth)
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
i-Minds Professional Stakeholders Qualitative Study | 24 weeks
  We will conduct semi-structured interviews and focus groups either by phone or online with up to 30 healthcare professionals who work within Child and Adolescent Mental Health Services, Sexual Assault Referral Centres or with an e-therapy provider. We will seek healthcare professionals' perspectives on the development of an online intervention designed to support young people who have experienced online sexual abuse (YP-OSA), including its advantages and disadvantages, how it compares with what services currently offer to YP-OSA, who it might benefit, what it should target, what will encourage or discourage YP to engage in the intervention, and how it could be scaled up and integrated sustainably within existing services. Data will be used to support the design of an online intervention for YP-OSA and the development of study information material and standard operating procedures of the subsequent feasibility study aimed at testing the intervention with YP-OSA.

CONTACTS AND LOCATIONS:
Locations (4):
- United Kingdom (4):
  - Greater Manchester Mental Health NHS Foundation Trust, Manchester, Lancashire
  - Manchester University Foundation Trust, Manchester, Lancashire
  - Pennine Care NHS Foundation Trust, Manchester, Lancashire
  - NHS Lothian, Edinburgh

IPD SHARING:
Plan to Share IPD: No
Qualitative research data will be shred within the research team but consent is not being sought to share data outside of the immediate research team